CLINICAL TRIAL: NCT02265016
Title: Regulation and Signaling of RBC-eNOS in Patients With Stable and Unstable Coronary Artery Disease
Brief Title: Regulation and Signaling of Red Blood Cell (RBC) Endothelial Nitric Oxide Synthase (eNOS) in Patients With Stable and Unstable Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator Prof. Dr. Malte Kelm, Heinrich-Heine University, Duesseldorf
Other Study IDs: RBC in CAD; 13-037 (Other: CTSU)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Endothelial NO-synthase
Keywords: coronary artery disease; acute coronary syndrome; angina pectoris; non-ST-segment elevation myocardial infarction; red blood cells; erythrocytes
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with CAD: Patients with stable coronary artery disease
- Patients with ACS: Patients with acute coronar syndrome, instable Angina pectoris and low-risk NSTEMI
- healthy control group: healthy control group without clinical apparent arteriosclerosis

SUMMARY:
The aim of this study is measurement of expression and activity of RBC eNOS in different clinical cohorts of patients with coronary artery disease and acute coronary syndrome and to investigate the importance of the NO-stimulated reaction cascade in terms of sGC and PKG.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* for ACS(acute coronary syndrome)-Group: angiographic coronary artery disease; acute coronary syndrome, defined by EITHER unstable angina pectoris with significant coronary stenosis (troponin negative, without significant ST-elevation) OR low-risk NSTEMI (Troponin positive, without significant ST-elevation)
* for stable CAD-Group: angiographic coronary artery disease; no acute coronary syndrome within the last 3 months
* healthy control group: No clinical or angiographical signs of apparent atherosclerosis

Exclusion Criteria:

* acute inflammation (CRP > 1 mg/dl, leukocyte > 11.000/µl)
* malignant diseases
* pregnancy
* medication with NO-donors ( e.g.isosorbide mononitrate, isosorbide dinitrate, glyceryl trinitrate, Molsidomin, Ranexa)
* patients with STEMI or high-risk NSTEMI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups:
  * ACS group (100 Patients)
  * stable CAD group (100 Patients)
  * healthy control group (100 Healthy Volunteers)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of red cell endothelial nitric oxide-synthase (eNOS)-expression and - activity | baseline, 3 hours and 3 month

SECONDARY OUTCOMES:
Deformability and stability of red blood cell membrane | baseline, 3 hours and 3 month
  by Laser assisted Optical Rotational Cell Analyzer (LORCA)
Microvascular function | baseline, 3 hours and 3 month
  Determination of microvascular function with Laser-Doppler Perfusion Imaging
Peripheral and central hemodynamic measurement | baseline, 3 hours and 3 month
Determination of arterial stiffness | baseline, 3 hours and 3 month
  Determination of arterial stiffness with pulse wave analysis during blood pressure measurement or echocardiography.
determination of flow-mediated dilation | baseline, 3 hours and 3 month
Determination of nitrate and nitrite in blood plasma and red blood cells (RBC) | baseline, 3 hours and 3 month
Determination of nitric oxide and cyclic guanosine monophosphate (cGMP) in blood plasma and in red blood cells | baseline, 3 hours and 3 month
Determination of endothelial microparticles | baseline, 3 hours and 3 month
Electrocardiogram | baseline, 3 hours and 3 month
Aging and turnover of red blood cells | baseline, 3 hours and 3 month
Redox status of red blood cells | baseline, 3 hours and 3 month
  Determination of redox status of red blood cells will be measured on free thiole with thioltracker and reactive oxygen species( ROS) by dihydrodichlorofluorescein
Aggregation of red blood cells | baseline, 3 hours and 3 month
  Determination of aggregation of red blood cells with LORCA
Platelet aggregometry | baseline, 3 hours and 3 month
Expression and function of soluble guanylyl cyclase (sGC) in red blood cells | baseline, 3 hours and 3 month
  measurement of enzyme expression and activity
Expression and activity of Protein Kinase G (PKG) | baseline, 3 hours and 3 month
  measurement of enzyme expression and activity
Determination of leucocyte populations and leucocyte function | baseline, 3 hours and 3 month
  flow-cytometry
Changes of tetrahydrobiopterin-metabolism | baseline, 3 hours and 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof. MD, Principal Investigator — Department of Cardiology, Pneumology and Angiology, University Hospital Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany